CLINICAL TRIAL: NCT01610219
Title: Lifestyle Modification for Type 2 Diabetes Prevention in Overweight Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 807106
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Modification for Diabetes Prevention (Active Comparator): Family based intervention utilizing Traffic Light Diet, self monitoring, parent behavioral skill training and tool kit of items promoting physical activity.
  Interventions: Behavioral: Lifestyle Modification for Type 2 Diabetes Prevention
- Nutrition and Physical Activity (Other): Family based intervention providing education on healthy eating and physical activity but no behavioral skills training, goal setting, self monitoring or physical activity toolkit.
  Interventions: Other: Nutrition and Physical Activity

INTERVENTIONS:
Behavioral: Lifestyle Modification for Type 2 Diabetes Prevention — Family based behavioral intervention utilizing Traffic Light Diet, self monitoring, goal setting, reinforcement and a tool kit containing physical activity-promoting items
  Arms: Lifestyle Modification for Diabetes Prevention
Other: Nutrition and Physical Activity — This family based education program provided information on physical activity and healthy eating for parents and children.
  Arms: Nutrition and Physical Activity

SUMMARY:
The number of youth with Type 2 diabetes (T2D) is rising in the population, which is a concerning public health trend. There has been little research testing ways to prevent the development of this disease in children who are at increased risk to develop T2D. This study tests a family treatment program that treats 4-8 year old children who are at risk for T2D because they are overweight and have a family history of the disease. Sixty at risk children and their parents were assigned to one of 2 treatment conditions. Half of the families (randomly determined) received an intensive family treatment program that trains parents in how to increase healthier foods choices and physical activity for themselves and their children using "behavior modification" strategies. Children receiving this treatment were allowed to taste new fruits and vegetables used a pedometer to record how far they walked every day, and were given a "tool box" of toys and interactive games which promoted physical activity. The other half of the families only received instruction about healthier choices, but received no behavioral modification strategies or physical activity promotion tools. Improvements in children's body weight, blood measures, and behavior patterns were measured after treatment ended (6 months) and then again after 12 months. The results may lead to a better understanding of how family members can positively influence young children's behaviors to help prevent T2D. The objective of proposed study was to test a family-based intervention designed to reduce excess body weight, improve metabolic and cardiovascular profile, and improve diet and physical activity levels in 4 - 8 year old youth who are "at risk" for T2D. This intervention was tested in a 2-arm randomized controlled clinical trial.

Primary Hypotheses:

1. Compared to children receiving NPA, children receiving LMDP will show greater reductions in excess body weight, greater improvements in metabolic and cardiovascular measures, improved diet, increased physical activity, and reduced television viewing.
2. Greater reductions in child excess body weight will be associated with greater improvements in metabolic and cardiovascular measures.

Secondary Hypotheses:

1. Compared to parents receiving the NPA intervention, parents receiving the LMDP intervention will show greater reductions in BMI.
2. Greater improvements in parent BMI will be associated with greater improvements in child body composition, metabolic and cardiovascular measures, and behavioral outcomes.
3. Compared to families receiving the NPA intervention, families receiving the LMDP intervention will show an increase in the number of fruits and vegetables and lower energy density foods stored at home.

DETAILED DESCRIPTION:
There is mounting concern about the development of Type 2 diabetes (T2D) in youth, especially in light of rising childhood obesity rates at younger ages. The health costs of T2D are notable both for the individual and society, and so interventions that can help prevent the development of T2D in early life are needed. Fortunately, there is promising evidence from the Diabetes Prevention Program (DPP) and other randomized trials with adults that the onset of T2D can be prevented through sustainable lifestyle changes. However, intervention programs have not been tested in young children who are "at risk" for developing the disease, even though this may be a critical period for obesity onset and for the formation of early eating and physical activity habits.

The primary aim of the proposed study was to test a family-based intervention that targets improvements in excess weight gain, metabolic and cardiovascular profile, and diet and physical activity in 4 - 8 year old children who are "at risk" for T2D. Specifically, 60 families were randomized either to one of two treatments: Lifestyle Modification for Diabetes Prevention (LMDP, N= 30) or Nutrition and Physical Activity Information (NPA, N= 30). The LMDP intervention trained families in behavioral strategies to increase parent and child intake of fruits, vegetables, and high fiber foods, to limit intake of energy-dense foods, and to increase daily physical activity. A physical activity "tool kit" for the home environment was provided to families. Supporting information about T2D and obesity, as well as nutrition and physical activity, also were provided. Besides the participating parent-child pair, other adult family members with T2D (eg, grandparents, aunts, uncles) were encouraged to participate. The LMDP activities were intended to reduce children's excess body weight and improve their metabolic and cardiovascular measures, to help prevent the onset of insulin resistance. The NPA intervention only received basic information on T2D and obesity, and nutrition and physical activity recommendations. Changes in child body composition, metabolic and cardiovascular measures, and behavioral outcomes were evaluated at 6 months (ie, end-of-treatment) and 12 months (ie, follow up). Changes in parent weight status and the home food environment were secondary outcomes and were assessed as potential mediators of child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-8 years old
* Age- and sex-specific BMI ≥95th percentile

Exclusion Criteria:

* Children with serious medical conditions
* Children who show signs of elevated psychopathology, as assessed by the Child Behavior Checklist (CBCL)
* Children of parents with significantly elevated psychiatric disorders

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline, 6 and 12 months
  Change in BMI will be measured from baseline to end of intervention (6 months) and and also from 6 months to 12 months.
BMI-z score | Baseline, 6 and 12 months
  Change in BMI-z score will be measured from baseline to end of treatment (6 months) and from 6 months to 12 months.
Percent overweight (% overweight) | Baseline, 6 and 12 months
  Change in percent overweight will be measured from baseline to end of treatment (6 months) and from 6 months to 12 months. Percent overweight is computed as a child's actual BMI minus the median BMI for a child of comparable sex and age, divided by 100.
Waist Circumference(cm) | Baseline, 6 and 12 months
  Change in waist circumference (cm) will be measured from baseline to end of treatment (6 months) and from end of treatment to 12 months.
Systolic Blood Pressure | Baseline, 6 and 12 months
  Change in systolic blood pressure (mm Hg) will be measured from baseline to end of treatment (6 months) and from end of treatment to 12 months.
Diastolic Blood Pressure (mm Hg) | Baseline, 6 and 12 months
  Change in diastolic blood pressure (mm Hg) will be measured from baseline to end of treatment (6 months) and from end of treatment to 12 months.
Pulse | Baseline, 6 and 12 months
  Change in resting pulse will be measured from baseline to end of treatment (6 months) and from end of treatment to 12 months.
Physical Activity | Baseline, 6 and 12 months
  Change in physical activity was measured from baseline to end of treatment (6 months) and from end of treatment to 12 months using an accelerometer. The accelerometer measured light, moderate and moderate-to-vigorous actity over 7 days.
Glucose | Baseline, 6 and 12 months
  Change in blood glucose levels were measured at baseline, 6 and 12 months.
Insulin | Baseline, 6 and 12 months
  Change in plasma insulin levels from baseline to end of treatment (6 months) and from 6 months to 12 months.
Change in HDL, LDL, Total Cholesterol and Triglycerides | Baseline, 6 and 12 months
  Change in lipid profile measures from baseline to end of treatment (6 months) and from 6 months to 12 months.
Change in Dietary Intake | Baseline, 6 and 12 months
  Change in energy (kcals/day), protein, carbohydrate, fat, cholesterol, saturated fat and fiber intake.

SECONDARY OUTCOMES:
Change in Parent BMI | Baseline, 6 and 12 months
  Change in parent BMI from baseline to end of treatment (6 months) and from 6 motnths to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Myles S Faith, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders/Perelman School of Medicine, Philadelphia, Pennsylvania, United States